CLINICAL TRIAL: NCT00795639
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Safety And Efficacy Study Of Sitaxsentan Sodium In Subjects With Pulmonary Arterial Hypertension
Brief Title: Sitaxsentan Efficacy And Safety Trial With A Randomized Prospective Assessment Of Adding Sildenafil (SR-PAAS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Safety Issue: The trial was prematurely terminated on Dec 9, 2010, due to safety concerns, specifically new emerging evidence of hepatic injury.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1321001
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2012-03-01 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Hypertension
Keywords: Sitaxsentan; endothelin receptor antagonist
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — sitaxsentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitaxsentan (Experimental): Monotherapy
  Interventions: Drug: Sitaxsentan
- Sitaxsentan Placebo (Placebo Comparator): Monotherapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitaxsentan — Sitaxsentan = 100 mg tablet administered orally, once daily
  Arms: Sitaxsentan
Drug: Placebo — Sitaxsentan Placebo = 1 tablet administered orally, once daily
  Other Names: Sitaxsentan Placebo
  Arms: Sitaxsentan Placebo

SUMMARY:
This protocol is for subjects with pulmonary arterial hypertension and is the first of 3 studies forming the Sitaxsentan efficacy and safety trial with Randomized Prospective Assessment of Adding Sildenafil (SR-PAAS) program.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of symptomatic pulmonary arterial hypertension (PAH) classified by one of the following: idiopathic arterial hypertension (IPAH), primary pulmonary hypertension (PPH), familial pulmonary arterial hypertension (FPAH) or pulmonary arterial hypertension (PAH) associated with connective tissue diseases. Has WHO functional class III symptoms.

Exclusion Criteria:

* Previous exposure to an endothelin receptor antagonist (ETRA) such as sitaxsentan, bosentan or ambrisentan.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (73):
- United States (31):
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Mather, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, Englewood, Colorado
  - Pfizer Investigational Site, Littleton, Colorado
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Weston, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Olathe, Kansas
  - Pfizer Investigational Site, Towson, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Islandia, New York
  - Pfizer Investigational Site, Stony Brook, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Lancaster, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Temple, Texas
  - Pfizer Investigational Site, Lynchburg, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Pfizer Investigational Site, Buenos Aires, Argentina
- Bulgaria (2):
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Veliko Tarnovo
- Pfizer Investigational Site, Temuco, Chile
- China (4):
  - Pfizer Investigational Site, Changsha, Hunan
  - Pfizer Investigational Site, Xi’an, Shanxi
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai
- Pfizer Investigational Site, Bogotá, Cundinamarca, Colombia
- Pfizer Investigational Site, Escazú, Provincia de San José, Costa Rica
- Pfizer Investigational Site, Prague, Czechia
- Dominican Republic (2):
  - Pfizer Investigational Site, Santo Domingo, República Dominicana
  - Pfizer Investigational Site, Santo Domingo, Santo Domingo Province
- Pfizer Investigational Site, Guatemala City, Departamento de Guatemala, Guatemala
- India (8):
  - Pfizer Investigational Site, Hyderabad, Andhera Pradesh
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Surat, Gujarat
  - Pfizer Investigational Site, Vadodara, Gujarat
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Coimbatore, Tamil Nadu
  - Pfizer Investigational Site, Madurai, Tamil Nadu
- Pfizer Investigational Site, George Town, Pulau Pinang, Malaysia
- Mexico (2):
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Monterrey, Nuevo León
- Pfizer Investigational Site, Lima, Peru
- Pfizer Investigational Site, Quezon City, Philippines
- Romania (2):
  - Pfizer Investigational Site, Cluj-Napoca, Romania
  - Pfizer Investigational Site, Iași
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Pfizer Investigational Site, Riyadh, Saudi Arabia
- Pfizer Investigational Site, Belgrade, Serbia
- Pfizer Investigational Site, Bratislava, Slovakia
- South Africa (4):
  - Pfizer Investigational Site, Cape Town, Western Cape
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Johannesburg
  - Pfizer Investigational Site, Stellenbosch
- Thailand (2):
  - Pfizer Investigational Site, Bangkoknoi, Bangkok
  - Pfizer Investigational Site, Bangkok
- Pfizer Investigational Site, Istanbul, Fatih, Turkey (Türkiye)
- Pfizer Investigational Site, Kyiv, Ukraine

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321001&StudyName=Sitaxsentan%20Efficacy%20And%20Safety%20Trial%20With%20A%20Randomized%20Prospective%20Assessment%20Of%20Adding%20Sildenafil%20%28SR-PAAS%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitaxsentan: Sitaxsentan 100 milligrams (mg) tablet orally once a day
- Placebo: Matching placebo tablet once a day
Period: Overall Study
Arm/Group | Sitaxsentan | Placebo
Started | 91 | 92
Randomized and Not Treated | 0 | 1
Completed | 70 | 66
Not Completed | 21 | 26
Not completed — Death | 1 | 6
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 5 | 2
Not completed — Other | 0 | 2
Not completed — Terminated by sponsor | 13 | 12
Not completed — Randomized and not treated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitaxsentan | Placebo | Total
Number analyzed (Participants) | 91 | 91 | 182
Age, Customized [Number; unit: participants]
  less than 18 years | 0 | 3 | 3
  18 to 44 years | 53 | 53 | 106
  45 to 64 years | 30 | 26 | 56
  greater than or equal to 65 years | 8 | 9 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 68 | 139
  Male | 20 | 23 | 43
World Health Organization (WHO) Functional Class [Number; unit: Participants] — WHO Pulmonary Arterial Hypertension (PAH) Functional Classification: I (no limitation on physical activity), II (slight limitation on ordinary physical activity), III (marked limitations on physical activity comfortable at rest) and IV (unable to carry out any physical activity without symptoms, dyspnea and fatigue present at rest).
  Participants
    Functional Class I | 0 | 0 | 0
    Functional Class II | 2 | 0 | 2
    Functional Class III | 88 | 87 | 175
    Functional Class IV | 0 | 0 | 0
    Functional Class Unknown | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Distance Walked During 6 Minute Walk Distance (6MWD) at Week 12
Description: 6 MWD was the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed. Continuous pulse oximetry was conducted during the test for safety. Change is Week 12 results minus baseline results.
Time Frame: Baseline/Day 1 and Week 12
Population: Intent to treat population (ITT): all participants who were randomized; missing value at Week 12 imputed with last non-missing value, including the non-missing value obtained at early termination based on last observation carried forward (LOCF)
Measure: Median (Full Range); unit: Meters (m)
Arm/Group | Sitaxsentan | Placebo
Number analyzed (Participants) | 91 | 92
Meters (m)
  Baseline | 343.0 [160 to 442] | 330.5 [169 to 456]
  Change at Week 12 | 13.0 [-349 to 105] | 3.0 [-338 to 104]
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; Test type: Superiority or Other; p = 0.0104, ANCOVA — Significance test performed using non-parametric analysis of covariance controlling for Baseline 6MWD and PAH etiology and PAH not secondary to a connective tissue disease (other); Mean Difference (Final Values) = 14, 95% CI 2-sided [3 to 26] — Missing value at Week 12 assigned as zero if the subject had a predefined clinical worsening event, otherwise, missing value at Week 12 imputed with the last non-missing 6MWD based on LOCF

2. Secondary Outcome: Number of Participants With Change From Baseline in World Health Organization (WHO) Functional Classification at Weeks 4, 8 and 12
Description: WHO functional classification for PAH ranges from Class I (no limitation in physical activity, no dyspnea with normal activity) to Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest). Improvement = reduction in functional class, deterioration = increase in functional class, no change = no change in functional class.
Time Frame: Baseline, Weeks 4, 8 and 12 or Early Termination (ET)
Population: ITT; N=number of participants with analyzable data; n=number of participants with analyzable data at the specific time point
Measure: Number; unit: participants
Arm/Group | Sitaxsentan | Placebo
Number analyzed (Participants) | 90 | 87
participants
  Week 4 - Improvement (n=90, 87) | 6 | 2
  Week 4 - No Change (n=90, 87) | 83 | 84
  Week 4 - Deterioration (n=90, 87) | 1 | 1
  Week 8 - Improvement (n=86, 81) | 13 | 6
  Week 8 - No Change (n=86, 81) | 72 | 73
  Week 8 - Deterioration (n=86, 81) | 1 | 2
  Week 12 - Improvement (n=80, 72) | 17 | 7
  Week 12 - No Change (n=80, 72) | 63 | 64
  Week 12 - Deterioration (n=80, 72) | 0 | 1
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; Week 12; Test type: Superiority or Other; p = 0.2908, Cochran-Mantel-Haenszel — Significance tests of WHO Functional Class performed using the Cochran-Mantel-Haenszel (CMH) test, stratified by Baseline 6MWD (less than 310 meters and greater than or equal to 310 meters) and PAH Etiology (Connective Tissue Disease and others); The CMH test used modified ridit scores, and the p-value corresponding to ANCOVA (row mean scores) statistics were used

3. Secondary Outcome: Time to Clinical Worsening (TTCW)
Description: TTCW defined as the number of days between first dose of study drug and the occurrence of a predefined clinical worsening event. Predefined clinical worsening events included: hospitalization for worsening PAH, on-study death, heart-lung or lung transplant, atrial septostomy or withdrawal due to the addition of any chronic medications for the treatment of worsening PAH.
Time Frame: Baseline, Weeks 4, 8 and 12 or ET
Population: ITT; N=number of participants with analyzable data
Measure: Median (Full Range); unit: days
Arm/Group | Sitaxsentan | Placebo
Number analyzed (Participants) | 91 | 91
days | NA [12 to 86] — Not Applicable (NA). TTCW not calculated unless at least 50 percent of participants in each treatment group had a clinical worsening event. | NA [3 to 73] — TTCW not calculated unless at least 50 percent of participants in each treatment group had a clinical worsening event.

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sitaxsentan | Placebo
Serious Adverse Events (participants affected / at risk) | 9/91 | 12/91
Other Adverse Events (participants affected / at risk) | 23/91 | 24/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (N=91) | Placebo (N=91)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Acute right ventricular failure (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Decreased activity (Psychiatric disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (N=91) | Placebo (N=91)
Vomiting (Gastrointestinal disorders) | 2 | 5
Chest pain (General disorders) | 2 | 3
Fatigue (General disorders) | 1 | 4
Oedema (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 5 | 8
Alanine aminotransferase increased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Dizziness (Nervous system disorders) | 5 | 2
Headache (Nervous system disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7

LIMITATIONS AND CAVEATS:
Study terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.